CLINICAL TRIAL: NCT05007457
Title: The Effectiveness of Respiratory Tele-rehabilitation After COVID-19 Pneumonia Related: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Angela Peghetti, Research Nurse, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ReF2002
Record Dates: First submitted 2021-04-12; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Failure; Sars-CoV-2; Covid19; ARDS; Interstitial Pneumonia; Respiratory Rehabilitation; Dyspnea; Quality of Life; Coronavirus Infections
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19; Lung Diseases, Interstitial; Dyspnea; Coronavirus Infections | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Partecipants, care providers and investigators are blinded only at the time of enrollment, subsequently they will learn about the group in which the partecipants were placed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): telerehabilitation
  Interventions: Other: Telerehabilitation
- Control group (Active Comparator): Standard treatment
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Patients belonging to the experimental group will receive the brochure and, weekly a telematic comparison will take place lasting about 30 minutes, with a physiotherapist to be asked questions. The physiotherapist will be able to evaluate and modify the training program based on the patient's response.
  The tele-rehabilitation sessions will take place: once / week for the first month, once every 2 weeks for the second month and from the third month from the third month the patient can contact the professionals in case of doubts or questions regarding the exercises he is taking place at home.

SUMMARY:
In recent months, more and more studies suggest tele-rehabilitation as a means to be exploited to reduce the risk of contagion.

The intent of our study is to verify the effectiveness of a tele-rehabilitation intervention through the application of a respiratory rehabilitation program supported by contact with physiotherapists, in patients with outcomes from SARS-CoV-2 infection discharged from the various medical departments and taken over by physiotherapists after physiatric evaluation.

Faced with the same rehabilitation program prescribed to all patients, the primary objective of our study is to detect whether patients supported by remote rehabilitation after hospitalization improve both adherence to the rehabilitation program and cardiorespiratory endurance and dyspnea symptoms assessed with the Six Minute Walking Test scale (6MWT). This test is validated for multiple pathologies, including idiopathic pulmonary fibrosis, the clinic of which could be comparable to the outcomes of coronavirus interstitial pneumonia as suggested by the literature.

The secondary objectives concern the assessment of the impact of physical exercise assisted by tele-rehabilitation detected through: the assessment of the quality of life (Saint George Respiratory Questionnaire );the assessment of autonomy in daily life activities (Barthel Index Dyspnea Scale), the evaluation of the variation in thoracic expansion and lung volumes (with COACH , an instrument for respiratory physiotherapy that measures the inspiratory volume in ml); the evaluation of muscle strength and endurance (One Minute Sit To Stand) ; the detection of dyspnea during the execution of the exercises (Modified Borg scale); the assessment of the functionality of the lower limbs (Short Physical Performance Battery)

DETAILED DESCRIPTION:
With regard to respiratory problems, there are still no precise data on the long-term consequences of pulmonary fibrosis and therefore related to the insufficient functioning of the lung. It is possible to hypothesize that these deficiencies can be treated with one specific respiratory rehabilitation aimed at reducing dyspnea and difficulty in practicing daily activities and moving around. In fact, the scientific literature indicates that respiratory rehabilitation improves the quality of life and exercise tolerance of patients with IPF (idiopathic Pulmonary Fibrosis), by reducing respiratory deficits, hypotrophy and muscle weakness, physical deconditioning. Respiratory rehabilitation means a "multidisciplinary intervention based on scientific evidence for patients with chronic respiratory disorders who are symptomatic and often have a reduced quality of life, in need of aerobic and respiratory muscle training, but also oxygen, nutritional, educational, psychological support as well as therapeutic education. For all these reasons we have decided to start our blinded, single-center randomized controlled study, the details of which will be specified later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID19;
* Respiratory failure in Sars-Cov2 pneumonia;
* ARDS in Sars-Cov2 pneumonia;
* Interstitial pneumonia from Sars-Cov2;
* Rankin scale ≥ 3/5 before enrollment (therefore at discharge);
* Patients in need of rehabilitation;
* Patients discharged from the hospital at their home;
* Patients with internet access;
* Owners and users of smartphones / tablets / PCs;
* Owners a pedal / stationary bike and oximeter.

Exclusion Criteria:

* Asymptomatic or paucisymptomatic patient;
* Institutionalized person;
* Unstable angina;
* Recent IMA;
* Life expectancy <12 months for other comorbidities (eg advanced cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-06-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walking Test (6MWT) | through study completion, an average of 1 year
  Six Minute Walking Test (6MWT) variation of more than 21.7 meters after 10 weeks of rehabilitation (the least clinically significant variation in patients with IPF - idiopathic pulmonary fibrosis - for the 6MWT is more than 21.7 meters after 6 months of rehabilitation)

SECONDARY OUTCOMES:
Improvement of daily living activities | through study completion, an average of 1 year
  Barthel Index Dispnea (BID)
Improvement of thoracic expansion and lung volumes | through study completion, an average of 1 year
  COACH (volume incentive used in respiratory rehabilitation)
Improvement of muscle strength and endurance | through study completion, an average of 1 year
  6 minute walking test (6MWT) One Minute Sit To Stand (1MSTS) Short Physical Peformance Battery (SPPB)
Improvement of the quality of life | through study completion, an average of 1 year
  St. George's Respiratory Questionnaire (SGRQ)
Improvement of dyspnea in the execution of life activities | through study completion, an average of 1 year
  Barthel Index Dispnea (BID)
Improvement of the functionality of the lower limbs | through study completion, an average of 1 year
  One Minute Sit To Stand (1MSTS) Short Physical Peformance Battery (SPPB)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Guerrieri, Director, Study Director — AOSP Bologna
Locations (1):
- Angela Peghetti, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Jiang J, Wang R, Fu H, Lu J, Yang M. Chest physiotherapy for pneumonia in adults. Cochrane Database Syst Rev. 2022 Sep 6;9(9):CD006338. doi: 10.1002/14651858.CD006338.pub4. PMID 36066373
- Available data/document: Study Protocol: Benedetta Isani — http://aosp.bo.it